CLINICAL TRIAL: NCT04185935
Title: Molecular Genetics Studies of Cancer Patients and Their Relatives
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 96144; NCI-2019-05695 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 96144 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2019-12-03; First posted 2019-12-04 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, eyebrow pluck, urine, tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-correlative (biospecimen collection): Participants may provide a sample of blood, a saliva sample, a sample of eyebrow plucks, a sample of urine, and/or stored tumor or healthy tissue.
  Interventions: Other: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Other: Biospecimen Collection — Provide a sample of blood, a saliva sample, a sample of eyebrow plucks, a sample of urine, and/or stored tumor or healthy tissue
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the genetic and behavioral factors that may contribute to the development of specific cancers and how these factors may affect the outcome of the disease in patients with a history of cancer and their relatives.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify rare cancer patients and families in whom the pattern of disease suggests a genetic susceptibility to cancer or other etiology suggestive of a carcinogenic exposure and to characterize the underlying predisposition.

II. To determine the contribution of heredity (genotype) and biomarkers to clinical outcome (phenotype, occurrence of new cancers, prognosis and quality of life) in subgroups of cancer patients with and without clinical high-risk features.

OUTLINE:

Patients may provide a sample of blood, a saliva sample, a sample of eyebrow plucks, a sample of urine, and/or stored tumor or healthy tissue.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must have a personal history of cancer and/or a family history of cancer suggestive of the presence of an inherited predisposition. This inherited predisposition might manifest as:

  * Young age cancer diagnosis
  * Multiple primary neoplasms in affected member
  * The presence of rare tumor types in the family
  * Congenital malformations
  * Any other family clustering of cancer
  * Any other cancer-predisposing genetic diseases/conditions
* Individuals may also be eligible by participation in the City of Hope Cancer Screening & Prevention Program Network (CSPPN) clinical service or on the basis of membership in a group known or suspected to have an increased risk of carrying a genetic alteration or of sustaining a particular exposure that would place that at increased risk of cancer. (Examples would include members of occupational cohorts like asbestos workers, individuals with multiple dysplastic nevi in the absence of a family history of cancer, and individuals descended from a particular tribe in the American Southwest who have an increased incidence of a rare genetic alteration associated with an increased risk of a specific cancer.)
* Individuals and families may be referred to us in a number of different ways. After initial contact is made with a individual or family by family studies personnel; an individual within the bloodline will be identified as the historian. There may be more than one historian within a family
* At least one historian must be wiling to provide information or access as needed to contact appropriate family members for documentation of cancer and for consent. An individual is considered to be eligible to participate if they criteria; contact with relatives is not always indicated
* Individuals who are under 18 are eligible for study if they meet the criteria. Consent for participation must be given by a legal guardian or parent
* Deceased patients may be included in the study. Public records, such as death certificates, can be used to confirm information from individuals or family members. If medical records are needed, consent for these records will be obtained from the deceased's next of kin. Next of kin refers to the following hierarchy of relatives; spouse, offspring, parents, and siblings. (Any further use of next of kin in this protocol should relate back to this hierarchy.) Archived tissue samples, such as pathology blocks or snap frozen tumor from a pathology department tumor bank (discard specimens) may be used for genetic research

Exclusion Criteria:

* A family may be ineligible for study if the historian will not allow access to anyone within the family and thus, the accuracy of the family history cannot be established

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with a family history of cancer
Sampling Method: Probability Sample
Enrollment: 999999 (Estimated)
Dates: Start 1997-04-18 (Actual); Primary Completion 2033-08-18 (Estimated); Study Completion 2033-08-18 (Estimated)

PRIMARY OUTCOMES:
Cancer risk assessment | Up to 10 years
Exploratory biomarkers for future studies | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gruber, MD, Principal Investigator — City of Hope Medical Center
Locations (42):
- United States (35):
  - Valleywise Comprehensive Health Center - Phoenix, Phoenix, Arizona
  - John Muir Medical Center-Concord Campus, Concord, California
  - City of Hope Medical Center, Duarte, California
  - Saint Jude Medical Center, Fullerton, California
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Lynn Regional Cancer Center - West, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Kootenai Cancer Center, Post Falls, Idaho
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Mercy Hospital, Cedar Rapids, Iowa
  - Suburban Hospital, Bethesda, Maryland
  - Frederick Oncology Hematology Associates, Frederick, Maryland
  - Steward Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Hunterdon Medical Center, Flemington, New Jersey
  - Lovelace Medical Center-Downtown, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Mount Kisco Medical Group at Northern Westchester Hospital, Mount Kisco, New York
  - Health Quest Medical Practice PC-Cardio Thoracic, Poughkeepsie, New York
  - Aultman Health Foundation, Canton, Ohio
  - Saint Charles Health System, Bend, Oregon
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Covenant Medical Center, Lubbock, Texas
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
- Colombia (2):
  - Clinica del Country, Bogotá, Cundinamarca
  - Instituto de Cancerologia Las Americas, Medellín
- Mexico (3):
  - University of Guadalajara, Guadalajara, Jalisco
  - Salvador Zubiran National Institute of Health Sciences and Nutrition, Mexico City, Tlalpan
  - Monterrey Institute of Technology-TecSalud, Nuevo León
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- University of Puerto Rico, San Juan, Puerto Rico